CLINICAL TRIAL: NCT04127500
Title: The Mechanism of Dexmedetomidine in Improving Delirium After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, HONG LIANG, Doctor, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20190823-04
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Dexmedetomidine; Delirium; Cardiac Surgery
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Experimental): use DEX
  Interventions: Drug: dexmedetomidine
- control group (No Intervention): use placebo

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine
  Arms: DEX group

SUMMARY:
The investigators aim to evaluate the roles of α7nAchR in the mechanisms of dexmedetomidine in improving delirium after cardiac surgery. The results of this study would lay the foundation for revealing the mechanisms of dexmedetomidine improving delirium after cardiac surgery and provide a new idea to the early treatment of delirium.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients underwent cardiac surgery
* age ≥ 60 years

Exclusion Criteria:

* Preoperative cognitive decline, mental illness,
* preoperative long-term use of hormone patients,
* preoperative alcohol dependence,
* patients with alcohol withdrawal symptoms

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
delirium incidence | 1 month
α7nAChR level | 7 days

SECONDARY OUTCOMES:
mechanical ventilation time | 7 days
ICU stay time | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No